CLINICAL TRIAL: NCT03860493
Title: Feasibility of the IC-Flow Device for Fluorescent Perfusion Evaluation During Open Surgical Procedures
Brief Title: Feasibility of the IC-Flow Device for Fluorescent Perfusion Evaluation During Feasibility of the IC-Flow Device
Acronym: IC-Flow
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: FLA 19-008
Record Dates: First submitted 2019-02-27; First posted 2019-03-04 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Skin Flap Necrosis; Perfusion; Complications
Keywords: organ perfusion; Fluorescence; icg
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Only patients who might benefit from intraoperative fluorescent tissue perfusion assessment according to the primary surgeon will be enrolled in the study. The patients will be screened and consent during their office visit with their surgeon at the Cleveland Clinic Foundation. Each surgeon will follow the standard Open surgical protocol of his/her subspecialty, and will comply with the following additional steps according to the type of surgery:
  Interventions: Procedure: Perfusion evaluation with indocyanine green

INTERVENTIONS:
Procedure: Perfusion evaluation with indocyanine green — 1. At least 10 minutes before surgery, will receive a weight-scaled dose of indocyanine green by IV and the time of administration and any adverse reactions will be recorded. The Surgeon/researcher will visualize and record the images given by the KARL STORZ VITOM II ICG System and the IC-Flow camera.
  3. The surgery will proceed as planned pre-operatively. The surgeon will conduct the surgery under white light and will categorize initial visualization of the organs.

SUMMARY:
1. Primary Objective:

   Demonstrate that the IC-Flow Imaging device with Indocyanine Green (ICG) is a feasible technique when visualizing and identifying perfusion of organs when compared to The KARL STORZ VITOM II ICG System during open reconstructive surgical procedures
2. Secondary Objective:

   1. Evaluate the mean Assessment of handling properties using The IC- Flow versus The VITOM II.
   2. Evaluate the mean Surgeon preference Level using The IC- Flow tower, The IC-Flow Hand-held device versus The VITOM II.

DETAILED DESCRIPTION:
Currently, there is no literature that supports the clinical application of the IC-Flow. However, we intend to perform this pilot study to determine safety and feasibility of said device in comparison to its homologue, FDA-approved VITOM II ICG System.

The device named The KARL STORZ VITOM II ICG System is an imaging system used in capturing and viewing fluorescent images. The system is FDA approved for all the indications that are going to be used in our study as well as the specialties involved It is composed of an open field multidirectional imaging arm and head, a light guide and a video processor/illuminator (FDA 510 (k) K171238, May 25, 2017).

As indicated by the Department of Health and Human Services from the FDA, the indications for use are the following: "The system is used in capturing and viewing fluorescence images for the visual assessment of blood flow as an adjunctive method for the evaluation of tissue perfusion, and related tissue-transfer circulation in tissue and free flaps used in plastic, micro- and reconstructive surgical procedures." And "The system is intended to provide fluorescence images for the visual assessment of blood flow in vessels and related tissue perfusion during gastrointestinal procedures." Based on the information provided by the FDA, the device has no direct nor indirect effect on patients. Furthermore, the device predicts a safe use and it's intended to provide imagery feedback alone.

There is few clinical trials which broadly exemplify the alternate applications of ICG fluorescence as a diagnostic tool for intraoperative anatomical identification, in terms of structure, perfusion, and tissue viability. No significant increase of risks or dye-associated complications had been reported.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders
2. Minimum age: 18 years old
3. Spoken and written command of the language spoken in the country's center
4. Ability to understand and follow the study procedures and sign the informed consent
5. open surgical porcedures

Exclusion Criteria:

1. Known allergies to iodides
2. Known history of coagulopathy
3. Women who are pregnant or breastfeeding, or for whom possibility of pregnancy was not ruled out

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will include patients aged 18-years old and above, selected for open reconstructive surgical procedures.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Perfusion with The KARL STORZ VITOM II ICG and IC-FLow System | 1 to 4 hours
  The vascular perfusion of the tissue studied will be analyzed using the infra red light after injection of indocyanine green (ICG) by using both the Karl Storz Vitom II and the IC-Flow systems.

SECONDARY OUTCOMES:
handling properties and surgeon preference level | 1 to 4 hours
  The images attained from the two systems (Vitom II vs. IC-Flow) will be evaluated. Also the handling properties of the two devices (ease to use, portability, set up, hardware, etc) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Lo Menzo, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dip FD, Asbun D, Rosales-Velderrain A, Lo Menzo E, Simpfendorfer CH, Szomstein S, Rosenthal RJ. Cost analysis and effectiveness comparing the routine use of intraoperative fluorescent cholangiography with fluoroscopic cholangiogram in patients undergoing laparoscopic cholecystectomy. Surg Endosc. 2014 Jun;28(6):1838-43. doi: 10.1007/s00464-013-3394-5. Epub 2014 Jan 11. PMID 24414461
- [Result] Alander JT, Kaartinen I, Laakso A, Patila T, Spillmann T, Tuchin VV, Venermo M, Valisuo P. A review of indocyanine green fluorescent imaging in surgery. Int J Biomed Imaging. 2012;2012:940585. doi: 10.1155/2012/940585. Epub 2012 Apr 22. PMID 22577366
- [Result] Choi M, Choi K, Ryu SW, Lee J, Choi C. Dynamic fluorescence imaging for multiparametric measurement of tumor vasculature. J Biomed Opt. 2011 Apr;16(4):046008. doi: 10.1117/1.3562956. PMID 21529077
- [Result] Kang Y, Choi M, Lee J, Koh GY, Kwon K, Choi C. Quantitative analysis of peripheral tissue perfusion using spatiotemporal molecular dynamics. PLoS One. 2009;4(1):e4275. doi: 10.1371/journal.pone.0004275. Epub 2009 Jan 26. PMID 19169354